CLINICAL TRIAL: NCT01115452
Title: A Proof of Principle Study Investigating the Effects of a Potassium Nitrate Solution in Reducing Dentinal Hypersensitivity
Brief Title: Efficacy of Potassium Nitrate Solution in Reducing Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z3770633
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Dentine Hypersensitivity
Keywords: potassium nitrate; tooth sensitivity; dentin sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5% KNO3 solution (Experimental): Participants to apply 5% potassium nitrate solution to a single sensitive tooth for two minutes, in each of the five day treatment period.
  Interventions: Drug: 5% Potassium nitrate
- 2.5% KNO3 solution (Experimental): Participants to apply 2.5% potassium nitrate solution to a single sensitive tooth for two minutes, in each of the five day treatment period.
  Interventions: Drug: 5% Potassium nitrate; Drug: 2.5% Potassium nitrate
- Sterile Water (Placebo Comparator): Participants to apply sterile water to a single sensitive tooth for two minutes, in each of the five day treatment period.
  Interventions: Other: Sterile water

INTERVENTIONS:
Drug: 5% Potassium nitrate — 5% potassium nitrate solution
  Arms: 2.5% KNO3 solution; 5% KNO3 solution
Drug: 2.5% Potassium nitrate — 2.5% potassium nitrate solution
  Arms: 2.5% KNO3 solution
Other: Sterile water — Sterile water
  Arms: Sterile Water

SUMMARY:
An exploratory study investigating the direct application of potassium nitrate (KNO3) solutions of different concentrations in reducing dentine hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of dentinal hypersensitivity lasting more than 6 months and a primary complaint of sensitive teeth
* Three teeth that can be isolated that meet all of the following criteria at the screening visit:
* Teeth showing signs of facial/cervical gingival recession and/or signs of erosion or abrasion. Study teeth must exhibit greater than or equal to 3 mm recession at the facial surface midpoint
* Teeth must be visually stain and calculus free
* Teeth having a gingival index score of less than or equal to 2
* Teeth with a clinical mobility less than or equal to 1
* Teeth that show signs of sensitivity, evaporative (air) sensitive teeth displaying a response of greater than or equal to 30 mm on a 100 mm VAS

Exclusion Criteria:

* Chronic disease or other condition that is associated with intermittent episodes of constant daily pain, such as arthritis, low back pain, etc.
* An condition or medication that causes xerostomia as determined by investigator
* Sensitive teeth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator
* Teeth with exposed dentine but with deep, defective or facial restorations
* Teeth used as abutments for fixed or removable partial dentures
* Teeth with full crowns, orthodontic bands, extensive caries or cracked enamel
* Sensitive teeth with contributing etiologies other than erosion, abrasion or recession of exposed dentine.
* Dental prophylaxis within 3 weeks of the screening visit
* Tongue or lip piercing or presence of dental implants
* Subjects not using the same brand of toothpaste for at least 4 months prior to the screening visit
* Subjects who have used desensitizing toothpaste during the 4 weeks before Treatment Visit 1
* Taking daily dose of medication which may interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquillizers, mood-altering drugs or anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- University Park Research Center (UPRC), Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site
Pre-assignment Details: Participants with at least three non-adjacent sensitive teeth were included in the study. Each participant received three treatments during each of the five days treatment. Treatments were randomly assigned to each of the three individual sensitive tooth.
Groups:
- 5% or 2.5% Potassium Nitrate Solution or Water: Investigator applied the participants with 5% potassium nitrate solution or 2.5% potassium nitrate solution or water to a single sensitive tooth for two minutes (mins), in each of the five day treatment period. This was a split-mouth design where three teeth were treated but each tooth had a different treatment.
Period: Overall Study
Arm/Group | 5% or 2.5% Potassium Nitrate Solution or Water
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 5
Region of Enrollment [Number; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Immediately Following Treatment on Day 5 Using a Visual Analog Scale (VAS) in 5% Potassium Nitrate Solution and 2.5% Potassium Nitrate Solution
Description: Response to a one second application of air from a standard dental unit syringe applied to the surface of hypersensitive tooth. After each stimuli participant rated the intensity of pain on a 100 millimeter VAS, on which 0 represented "no pain" and 100 represented the" worst pain imaginable". Change from baseline was calculated as mean score at the given time point minus mean score at baseline.
Time Frame: Baseline and immediately after treatment on Day 5
Population: Intent to treat (ITT) population: All participants who were randomized, receive at least one dose of treatment, and had at least one post baseline efficacy evaluation. There was no imputation for missing data. Analysis population was less than the randomized population because 2 participants had one tooth which was not treated
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- 5% Potassium Nitrate Solution: Investigator applied the participants with 5% potassium nitrate solution to a single sensitive tooth for two mins, in each of the five day treatment period. This was a split-mouth design where three teeth were treated but each tooth had a different treatment.
- 2.5% Potassium Nitrate Solution: Investigator applied the participants with 2.5% potassium nitrate solution to a single sensitive tooth for two mins, in each of the five day treatment period. This was a split-mouth design where three teeth were treated but each tooth had a different treatment
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution
Number analyzed (Participants) | 30 | 30
units on a scale | -24.36 [-31.56 to -17.16] | -24.04 [-31.24 to -16.84]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis was no difference between treatments; Test type: Superiority or Other; p = 0.9347, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Treatment group, treatment application site and assessment time were fixed factors, baseline VAS was a covariate and participant was a random factor; Adjusted mean difference = -0.32, 95% CI 2-sided [-8.14 to 7.50] — Difference was calculated as adjusted mean change from baseline in 5% potassium nitrate solution minus 2.5% potassium nitrate solution. Negative difference favored 5% potassium nitrate solution

2. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Immediately Following Treatment on Day 1 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and immediately after treatment on Day 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Water: Investigator applied the participants with sterile water to a single sensitive tooth for two mins, in each of the five day treatment period. This was a split-mouth design where three teeth were treated but each tooth had a different treatment.
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -8.18 [-15.35 to -1.02] | -8.20 [-15.37 to -1.04] | -12.08 [-19.31 to -4.86]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9963, ANCOVA — Treatment group, treatment application site and assessment time were fixed factors, baseline VAS was a covariate and participant was a random factor; No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Adjusted mean difference = 0.02, 95% CI 2-sided [-8.20 to 8.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.3582, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 3.90, 95% CI 2-sided [-4.45 to 12.25] — Difference was calculated as adjusted mean change from baseline in 5% potassium nitrate solution minus water. Negative difference favored 5% potassium nitrate solution
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.3600, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 3.88, 95% CI 2-sided [-4.46 to 12.22] — Difference was calculated as adjusted mean change from baseline in 2.5% potassium nitrate solution minus water. Negative difference favored 2.5% potassium nitrate solution

3. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 10 Mins Post Treatment on Day 1 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 10 mins post treatment on Day 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -13.38 [-20.55 to -6.22] | -12.47 [-19.63 to -5.31] | -12.48 [-19.71 to -5.26]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8265, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.91, 95% CI 2-sided [-9.13 to 7.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8314, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.90, 95% CI 2-sided [-9.25 to 7.45] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9978, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.01, 95% CI 2-sided [-8.33 to 8.35] — [estimate comment as in outcome 2, analysis 3]

4. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 20 Mins Post Treatment on Day 1 Using a VAS.
Description: as for outcome 1
Time Frame: Baseline and 20 mins post treatment on Day 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -17.42 [-24.58 to -10.25] | -21.64 [-28.80 to -14.47] | -16.15 [-23.37 to -8.92]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.3122, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 4.22, 95% CI 2-sided [-4.00 to 12.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7646, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.27, 95% CI 2-sided [-9.62 to 7.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.1957, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -5.49, 95% CI [-13.83 to 2.85] — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Following Treatment on Day 2 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and immediately after treatment on Day 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -11.66 [-19.03 to -4.29] | -10.31 [-17.67 to -2.94] | -12.32 [-19.76 to -4.89]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7472, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.35, 95% CI 2-sided [-9.62 to 6.92] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8767, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.66, 95% CI [-7.75 to 9.08] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6367, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 2.01, 95% CI [-6.39 to 10.42] — [estimate comment as in outcome 2, analysis 3]

6. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 10 Mins Post Treatment on Day 2 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 10 mins post treatment on Day 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -18.09 [-25.46 to -10.72] | -16.14 [-23.51 to -8.77] | -18.52 [-25.96 to -11.09]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6417, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.95, 95% CI 2-sided [-10.22 to 6.32] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9200, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.43, 95% CI 2-sided [-7.99 to 8.85] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.5766, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 2.38, 95% CI [-6.02 to 10.78] — [estimate comment as in outcome 2, analysis 3]

7. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 20 Mins Post Treatment on Day 2 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 20 mins post treatment on Day 2
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -20.39 [-27.76 to -13.02] | -16.81 [-24.17 to -9.44] | -18.69 [-26.12 to -11.25]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.3930, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -3.58, 95% CI 2-sided [-11.65 to 4.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6896, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.70, 95% CI 2-sided [-10.12 to 6.71] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6591, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjustes mean difference = 1.88, 95% CI 2-sided [-6.52 to 10.28] — [estimate comment as in outcome 2, analysis 3]

8. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Immediately Following Treatment on Day 3 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and immediately after treatment on Day 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -16.66 [-24.48 to -8.84] | -14.58 [-22.40 to -6.76] | -14.90 [-22.79 to -7.00]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6301, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -2.08, 95% CI [-10.60 to 6.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6888, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.76, 95% CI 2-sided [-10.46 to 6.93] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9428, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.32, 95% CI 2-sided [-8.37 to 9.00] — [estimate comment as in outcome 2, analysis 3]

9. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 10 Mins Post Treatment on Day 3 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 10 mins post treatment on Day 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -23.29 [-31.12 to -15.47] | -20.71 [-28.53 to -12.89] | -21.20 [-29.09 to -13.30]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.5504, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -2.58, 95% CI 2-sided [-11.10 to 5.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6340, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -2.10, 95% CI 2-sided [-10.80 to 6.60] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9127, ANCOVA; No adjustment for multiple comparisons were made as the primary comparison was pre-defined; Adjusted mean difference = 0.48, 95% CI 2-sided [-8.20 to 9.16] — [estimate comment as in outcome 2, analysis 3]

10. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 20 Mins Post Treatment on Day 3 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 20 mins post treatment on Day 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -24.86 [-32.68 to -17.04] | -22.71 [-30.53 to -14.89] | -25.46 [-33.36 to -17.57]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.6192, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -2.15, 95% CI 2-sided [-10.67 to 6.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8912, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.60, 95% CI 2-sided [-8.10 to 9.30] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.5321, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 2.75, 95% CI 2-sided [-5.93 to 11.43] — [estimate comment as in outcome 2, analysis 3]

11. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Following Treatment on Day 4 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and immediately after treatment on Day 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -21.89 [-29.26 to -14.52] | -18.52 [-25.89 to -11.15] | -22.63 [-30.08 to -15.19]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.4055, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -3.37, 95% CI 2-sided [-11.37 to 4.63] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8573, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.74, 95% CI 2-sided [-7.42 to 8.91] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.3193, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 4.12, 95% CI 2-sided [-4.03 to 12.27] — [estimate comment as in outcome 2, analysis 3]

12. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 10 Mins Post Treatment on Day 4 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 10 mins post treatment on Day 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -21.09 [-28.46 to -13.72] | -24.32 [-31.69 to -16.95] | -22.13 [-29.58 to -14.69]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.4264, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 3.23, 95% CI [-4.77 to 11.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8008, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 1.04, 95% CI 2-sided [-7.42 to 9.21] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.5969, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -2.18, 95% CI 2-sided [-10.33 to 5.97] — [estimate comment as in outcome 2, analysis 3]

13. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli 20 Mins Post Treatment on Day 4 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 20 mins post treatment on Day 4
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -27.92 [-35.30 to -20.55] | -22.78 [-30.15 to -15.41] | -27.53 [-34.98 to -20.09]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.2059, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -5.14, 95% CI 2-sided [-13.14 to 2.86] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9248, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.39, 95% CI 2-sided [-8.56 to 7.77] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.2508, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 4.75, 95% CI 2-sided [-3.40 to 12.90] — [estimate comment as in outcome 2, analysis 3]

14. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli Immediately Following Treatment on Day 5 Using a VAS in 5% Potassium Nitrate Solution and Water; 2.5% Potassiun Nitrate Solution and Water
Description: as for outcome 1
Time Frame: Baseline and immediately after treatment on Day 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -24.36 [-31.56 to -17.16] | -24.04 [-31.24 to -16.84] | -25.48 [-32.75 to -18.21]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7822, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 1.12, 95% CI 2-sided [-6.86 to 9.10] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7208, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 1.44, 95% CI 2-sided [-6.52 to 9.41] — [estimate comment as in outcome 2, analysis 3]

15. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 10 Mins Post Treatment on Day 5 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 10 mins post treatment on Day 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -27.83 [-35.03 to -20.63] | -26.47 [-33.67 to -19.27] | -28.88 [-36.15 to -21.61]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7318, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -1.36, 95% CI 2-sided [-9.18 to 6.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.7949, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 1.05, 95% CI 2-sided [-6.93 to 9.03] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.5507, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 2.41, 95% CI 2-sided [-5.56 to 10.37] — [estimate comment as in outcome 2, analysis 3]

16. Secondary Outcome: Between Treatment Comparison of the Adjusted Mean Change From Baseline of Response to Evaporative (Air) Stimuli at 20 Mins Post Treatment on Day 5 Using a VAS
Description: as for outcome 1
Time Frame: Baseline and 20 mins post treatment on Day 5
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 5% Potassium Nitrate Solution | 2.5% Potassium Nitrate Solution | Water
Number analyzed (Participants) | 30 | 30 | 30
units on a scale | -30.93 [-38.13 to -23.73] | -30.20 [-37.40 to -23.01] | -30.78 [-38.05 to -23.51]
Statistical Analysis 1: Comparison: 5% Potassium Nitrate Solution vs 2.5% Potassium Nitrate Solution; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8549, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.72, 95% CI 2-sided [-8.54 to 7.10] — Investigator applied the participants with 5% potassium nitrate solution on each of the three individual sensitive tooth for two minutes (mins), in each of the five day treatment period
Statistical Analysis 2: Comparison: 5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.9705, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.15, 95% CI 2-sided [-8.13 to 7.83] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: 2.5% Potassium Nitrate Solution vs Water; Null hypothesis is no difference between treatments; Test type: Superiority or Other; p = 0.8867, ANCOVA — No adjustment for multiple comparisons were made as the primary comparison was pre-defined; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = 0.57, 95% CI 2-sided [-7.39 to 8.54] — [estimate comment as in outcome 2, analysis 3]

ADVERSE EVENTS:
Time Frame: Baseline through 5 days post administration of last treatment
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.